CLINICAL TRIAL: NCT01958723
Title: Problem Specific Templates for Electronic Hospital Documentation
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 201300232
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Quality/Accuracy of Physician Documentation; Efficiency of Physician Documentation
Keywords: Problem Specific Template; Physician Documentation; Electronic Medical Record Documentation
MeSH Terms: interventions — Hospitalists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalists: Introduction of Problem Specific Templates
  Interventions: Other: Hospitalists

INTERVENTIONS:
Other: Hospitalists — Introduction of Problem Specific Templates

SUMMARY:
The emergence of electronic documentation has led to multiple new challenges for physicians. Despite positive expectations, many physicians have received electronic health systems with mixed results. Review of current literature has identified the following reasons for concern: increased time required for documentation, deteriorating quality of notes, mindless use of copy-and-paste functions, and fragmentation of clinical work from poorly designed computing workflows. The study of template use has not been done in a large scale or with clear outcome measurements. The purpose of this study is to examine the effects of Problem Specific Templates on quality, accuracy, and efficiency of physician documentation practices.

DETAILED DESCRIPTION:
This is a prospective cohort study, which will examine the effects of Problem Specific Templates on quality, accuracy, and efficiency of physician documentation practices. The Hospitalist physicians will be the subjects. All physicians of the Hospital Medicine Service will be invited to participate. For the intervention, participating Hospitalists will be trained on the use of templates for 20 common hospital problems. Once trained, the Hospitalists will be asked to use these templates for a one-month period. Pre-intervention and post-intervention medical records will be compared using chart reviews, validated document assessment instruments, physician surveys, and electronic medical record time auditing.

ELIGIBILITY:
Inclusion Criteria:

* Physicians: All physicians of the Hospital Medicine Service will be invited to participate

Exclusion Criteria:

* Any invited physicians who refuse to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians of the Hospital Medicine Service
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quality and Accuracy of Physician Documentation Practices (as measured through chart review) | 1 year
Efficiency of Physician Documentation Practices (as measured through the electronic medical record auditing function) | 1 year

SECONDARY OUTCOMES:
Frequency of Physician Use of Problem Specific Templates (as measured through chart review) | 1 year
Physician Assessment of Note-Documenting and Electronic Medical Record (as measured through Physician Questionnaire) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Raj Mehta, M.D., Principal Investigator — University of Florida; Robert Leverence, M.D., Study Chair — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States